CLINICAL TRIAL: NCT04527536
Title: Research of Diagnostic Value of Fecal miRNA and Intestinal Flora in Infants With BMJ
Brief Title: Research of Diagnostic Value for BMJ Infants
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiFMIH-2020-084
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- early-set BMJ group: Infants were admitted to our hospital at 4-7 days of age and were followed up to 28 days. Other pathological jaundice factors were excluded.Those who met the criteria were the early-onset BMJ group.
  Interventions: Diagnostic Test: Neonatal hyperbilirubinemia
- late-onset BMJ group: Infants were admitted to our hospital after 7 days of age and were followed up to 28-42 days or until the jaundice disappeared. Other pathological jaundice factors were excluded..Those who met the criteria were late-onset BMJ
  Interventions: Diagnostic Test: Neonatal hyperbilirubinemia
- healthy control: During the same period, the healthy newborns who were born in the obstetrics department of our hospital. These newborns were mainly breastfed or breastfed, and grew well. They were enrolled at 7-14 days of age and were followed up to 28-42 days without pathological jaundice.
  Interventions: Diagnostic Test: Neonatal hyperbilirubinemia

INTERVENTIONS:
Diagnostic Test: Neonatal hyperbilirubinemia — Neonatal hyperbilirubinemia：The total serum bilirubin exceeds the 95th percentile of the Bhutani neonatal hourly bilirubin nomogram.

SUMMARY:
Breast milk jaundice (BMJ) is the main cause of neonatal hyperbilirubinemia. Excessive serum unconjugated bilirubin level will not only cause the interruption or early termination of breastfeeding, but also cause kernicterus. Which can cause long-term dysfunction in infants. But for a long time, BMJ diagnosis has relied on clinical exclusive methods, lack of objective and reliable laboratory indicators. Which leads to misdiag. This project is a single-center, prospective nested case-control study. It is planned to establish a neonatal BMJ cohort. According to the admission criteria, 100 cases of early-onset BMJ and late-onset BMJ will be completed, and 100 healthy controls collected during the same period. , Compare the detection results of fecal miRNA and intestinal flora of the two groups of BMJ children and healthy controls, draw the ROC curve of the joint diagnosis, conduct research on the combined diagnostic value of fecal miRNA and intestinal flora analysis, and try to find the feasibility and practical value of diagnostic markers for feces in infants with BMJ.

DETAILED DESCRIPTION:
This project is a single-center, prospective nested case-control study to investigate feasibility and practical value of diagnostic markers in infants with BMJ.

According to the admission criteria, 100 cases of early-onset BMJ, 100 late-onset BMJ and 100 healthy controls will be selected. Their feces, peripheral venous blood and mothers' breast milk were collected for further testing. Compare the detection results of fecal miRNA and intestinal flora of the two groups of BMJ children and healthy controls, draw the ROC curve of the joint diagnosis, conduct research on the combined diagnostic value of fecal miRNA and intestinal flora analysis.

This study is to find the objective and reliable laboratory indicators to diagnose BMJ.

ELIGIBILITY:
Inclusion Criteria:

* All the following conditions must be met

  1. Term newborns admitted to hospital with "neonatal hyperbilirubinemia"
  2. Exclusive breastfeeding or mainly breastfeeding
  3. Exclude perinatal infection, G-6P-D deficiency, homoimmune hemolysis, polycythemia, scalp hematoma, intracranial hemorrhage, cholestasis, hypoglycemia, hypothyroidism, hypothermia, neonatal asphyxia, fetus Pathological jaundice factors such as delayed stool excretion.

Exclusion Criteria:

* As long as any one of the following conditions should be excluded

  1. During the follow-up period, breastfeeding was terminated or the daily milk powder intake exceeded 200 ml.
  2. Other pathological jaundice was diagnosed during the follow-up period.
  3. Take probiotics during the sampling period.
  4. The guardian asked to withdraw from the study halfway.

Ages: 4 Days to 42 Days | Sex: All
Age Groups: Child
Study Population: Newborn babies born from research start who diagnosed neonatal hyperbilirubinemia and healthy newborns
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Analysis of breast milk exosomes miRNA | 2021.10.01-2022.09.30
  Analysis of breast milk exosomes miRNA
Analysis of newborn feces miRNA and intestinal flora analysis | 2021.10.01-2022.09.30
  Analysis of newborn feces miRNA and intestinal flora analysis
UGT1A1 test in newborn blood | 2021.10.01-2022.09.30
  UGT1A1 test in newborn blood

CONTACTS AND LOCATIONS:
Overall Officials: Jing Li, Doctorate, Principal Investigator — Shanghai First Maternity and Infant Hospital